CLINICAL TRIAL: NCT04179955
Title: Intraoperative Costs and Patient Perceptions in Sacrocolpopexy for Prolapse
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emanuel Trabuco, Associate Professor of Obstetrics and Gynecology, Mayo Clinic
Other Study IDs: 19-005064
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Robotic sacrocolpopexy (a procedure for female pelvic organ prolapse) has been demonstrated to have equivalent surgical outcomes to open abdominal sacrocolpopexy and has been previously deemed more cost effective due to the longer hospital course following open procedures. The total cost of these procedures, including all costs of hospitalization as well as costs associated with the 30 days following surgery have previously been evaluated by the investigators. However, previous research is lacking in both the specific cost components that contribute to intraoperative cost of surgery as well as the patient perceived outcomes following these two procedures. This project aims to evaluate the marginal costs of surgery and to survey sacrocolpopexy patients to evaluate their satisfaction with outcomes and surgical scars.

DETAILED DESCRIPTION:
Abdominal sacrocolpopexy (ASC) is the gold standard operation to treat pelvic organ prolapse. The open approach has been associated with prolonged hospital stay and higher peri-operative morbidity, leading many providers to prefer a robotic approach. Even though robotic ASC overcomes many of the technical hurdles associated with laparoscopy, it is expensive, and it achieves cost effectiveness compared to open only because of large discrepancies in length of stay. Preliminary data at our institution suggests that with the introduction of ERAS, decreases in hospital stay after abdominal surgery have driven down the discrepancy in length of stay between open (1.8 days) and robotic (1.4 days) ASC. Previous analysis accounted for differences in OR time as well as postoperative stay. However, this cost data is obtained from data on billed charges rather than a summation of actual costs sustained; data on specific incurred costs is scant in the literature. Robotic surgery requires equipment and resources which also increase the price of the procedure. Specifically, Da Vinci robots are priced at $1.4 million, require $120,000 in annual maintenance contracts, and the cost of disposable instruments can reach $2000 per case. Instruments and disposable materials, while contracted at Mayo, do have published prices that may be used to better quantify intraoperative procedural costs.

In addition to questions about the cost effectiveness of robotic versus abdominal sacrocolpopexy, data on patient satisfaction comparing the two procedures is minimal. While abdominal and robotic approaches have similar efficacy, patient perceived equivalence has been largely assumed. Additionally, the literature frequently lists improved cosmesis as a benefit to robotic surgery, yet the studies on scar satisfaction between the two approaches are lacking.

Hypothesis: Intraoperative costs of abdominal sacrocolpopexy are significantly less than those in the robotic approach. However, patients who undergo robotic sacrocolpopexy have improved scar satisfaction and equivalent perceived surgical satisfaction.

This is a prospective cohort study of intraoperative time and materials in open versus robotic ASC.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Undergoing abdominal or robotic sacrocolpopexy with or without posterior vaginal repairs
* Willing and able to provide signed informed research consent
* Concurrent and prior hysterectomy

Exclusion Criteria:

* Repeat sacrocolpopexy
* Concurrent sling procedure
* Concurrent Pouch of Douglas repairs
* Concurrent anterior vaginal wall repairs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only as this involves surgery for pelvic organ prolapse.
Study Population: Adult females undergoing sacrocolpopexy at Mayo Clinic Rochester
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative cost of surgery | SIx weeks postop
  Cost of surgery will be ascertained by summing marginal costs of surgery, including operative and anesthesia time, instruments and medications
Patient Scar Assessment | Six weeks postop
  Patient satisfaction with their surgical scars from sacrocolpopexy will be assessed via the Patient Scar Assessment Survey (POSAS). This validated scar assessment scale ranges from 6 to 60, with higher scores indicating worse scar aesthetics and symptoms.

SECONDARY OUTCOMES:
Surgical satisfaction | Six weeks postop
  Patient satisfaction with surgery will be assessed via the Surgical Satisfaction Questionnaire(SSQ-8), a validated survey for surgical satisfaction. Scores range from 0 to 100, with higher scores denoting better surgical satisfaction.
Surgical satisfaction | Six months postop
  Patient satisfaction with surgery will be assessed via the Surgical Satisfaction Questionnaire(SSQ-8), a validated survey for surgical satisfaction. Scores range from 0 to 100, with higher scores denoting better surgical satisfaction.
Urinary symptoms | Six weeks postop
  Patient urinary symptoms will be compared preoperatively with postoperative scores via the International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI), a validated survey for female urinary symptoms. Scores range from 0 to 21, with higher scores indicating more urinary distress/dysfunction.
Urinary symptoms | Six months postop
  Patient urinary symptoms will be compared preoperatively with postoperative scores via the International Consultation on Incontinence Questionnaire Urinary Incontinence Short Form (ICIQ-UI), a validated survey for female urinary symptoms. Scores range from 0 to 21, with higher scores indicating more urinary distress/dysfunction.
Sexual function | Six months postop
  Patient sexual function will be compared preoperatively with postoperative scores via the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12), a survey for female sexual function. Scores range from 0 to 48, with higher scores indicating better sexual function.
Patient Scar Assessment | Six months postop
  Patient satisfaction with their surgical scars from sacrocolpopexy will be assessed via the Patient Scar Assessment Survey (POSAS). This validated scar assessment scale ranges from 6 to 60, with higher scores indicating worse scar aesthetics and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel C Trabuco, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No